CLINICAL TRIAL: NCT00997126
Title: Propofol Versus Alfentanil Versus Nitrous Oxide for Moderate Procedural Sedation in the Emergency Department
Brief Title: Propofol Versus Alfentanil Versus Nitrous Oxide for Moderate Procedural Sedation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hennepin Healthcare Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MMRF093030
Record Dates: First submitted 2009-10-12; First posted 2009-10-19 (Estimated); Results first posted 2017-01-27 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2016-12

CONDITIONS: Sedation
Keywords: propofol; alfentanil; nitrous oxide; moderate procedural sedation; Moderate Procedural Sedation in the Emergency Department
MeSH Terms: interventions — Propofol; Alfentanil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Propofol (Active Comparator): Propofol 1m g/kg IV followed by 0.5 mg/kg IV prn sedation
  Interventions: Drug: Propofol
- Alfentanil (Active Comparator): Sedation using alfentanil 10 ug/kg followed by 5 ug/kg prn sedation
  Interventions: Drug: Alfentanil

INTERVENTIONS:
Drug: Propofol — Propofol 1 mg/kg IV followed by 0.5 mg/kg prn sedation
  Arms: Propofol
Drug: Alfentanil — Alfentanil 10 ug/kg IV followed by 5 ug/kg prn sedation
  Arms: Alfentanil

SUMMARY:
This is a clinical trial of propofol and alfentanil as agents for moderated procedural sedation in patients undergoing sedation in the emergency department (ED).

DETAILED DESCRIPTION:
This was initially going to be a trial of propofol vs alfentanil vs nitrous oxide, but our use of nitrous oxide was discontinued before the trial began and the trial was conducted with only two arms

ELIGIBILITY:
Inclusion Criteria:

* Adults undergoing moderate procedural sedation in the Emergency Department

Exclusion Criteria:

* Age <18 years
* Pregnancy
* Intoxication
* Cannot give informed consent
* Allergy to any of the three study medications
* ASA physical status score > 2
* Patients who require deep procedural sedation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2009-10; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James R Miner, MD, Principal Investigator — Hennepin Healthcare Research Institute
Locations (1):
- Hennepin County Medical Center, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Propofol | Alfentanil
Started | 63 | 63
Completed | 56 | 52
Not Completed | 7 | 11
Not completed — Physician Decision | 7 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Propofol | Alfentanil | Total
Number analyzed (Participants) | 56 | 52 | 108
Age, Continuous [Median (Full Range); unit: years] | 36 [18 to 64] | 32 [18 to 82] | 34 [18 to 82]
Gender [Count of Participants; unit: Participants]
  Female | 31 | 23 | 54
  Male | 25 | 29 | 54

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Sub-clinical Respiratory Depression and Clinical Events Associated With Respiratory Depression During the Sedation Procedure
Time Frame: From one minute prior to start of procedure until the patient has returned to baseline mental status after the conclusion of the sedation procedure (~3-60 minutes depending on procedure duration)
Measure: Number; unit: participants
Arm/Group | Propofol | Alfentanil
Number analyzed (Participants) | 56 | 52
participants | 11 | 12

2. Secondary Outcome: Time to Return of Baseline Mental Status From Start of Procedure in Minutes
Time Frame: Single time point after completion of sedation procedure, measured from start of procedure until the patient returns to baseline mental status up to 24 hours
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Propofol | Alfentanil
Number analyzed (Participants) | 56 | 52
minutes | 13 [9 to 17] | 13 [10 to 17]

3. Secondary Outcome: Depth of Sedation Measured Using the OAAS Scale
Description: Observers Assesment of Alertness Scale, 5 responds normally to voice, 4 lethargic response to voice, 3 responds only to loud voice or light touch, 2 responds only to mild prodding or shaking, 1 responds only to painful stimuli, 0 no response to painful stimuli
Time Frame: Single measurement during sedation procedure
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Propofol | Alfentanil
Number analyzed (Participants) | 56 | 52
units on a scale | 2 [1 to 3] | 3 [2 to 4]

4. Secondary Outcome: Patient Reported Pain
Time Frame: Single measurement immediately after patient returns to baseline mental status after sedation procedure
Measure: Number; unit: participants
Arm/Group | Propofol | Alfentanil
Number analyzed (Participants) | 56 | 52
participants | 7 | 25

5. Secondary Outcome: Patient Reported Recall of the Procedure
Time Frame: Single measurement immediately after patient returns to baseline mental status after sedation procedure
Measure: Number; unit: participants
Arm/Group | Propofol | Alfentanil
Number analyzed (Participants) | 56 | 52
participants | 13 | 39
Statistical Analysis 1: Comparison: Propofol vs Alfentanil; Test type: Superiority or Other; p = 0.657, Chi-squared

ADVERSE EVENTS:
Time Frame: From 1 minute prior to the procedure until the patient returned to baseline mental status
Arm/Group | Propofol | Alfentanil
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/52
Other Adverse Events (participants affected / at risk) | 25/56 | 29/52
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Propofol (N=56) | Alfentanil (N=52)
any airway or respiratory adverse event (Respiratory, thoracic and mediastinal disorders) | 25 (30) | 29 (35) — interventions during the procedure associated with respiratory depression, or change in ventilation including an oxygen sat <93% or apnea >6 seconds

LIMITATIONS AND CAVEATS:
our capability of administering nitrous oxide was diminished as the trial was started, and the trial was conducted using on the propofol and alfentanil arms.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No